CLINICAL TRIAL: NCT01446783
Title: IGF-I Stimulation of Collagen Synthesis in Ehlers-Danlos Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Rie Harboe Nielsen, Principal Investigator, Bispebjerg Hospital
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: H-1-2011-010
Record Dates: First submitted 2011-09-27; First posted 2011-10-05 (Estimated); Last update posted 2012-11-20 (Estimated); Status verified 2012-11

CONDITIONS: Ehlers-Danlos Syndrome, Classic
Keywords: COL5A1; Collagen disorders; IGF-I; Collagen synthesis
MeSH Terms: conditions — Ehlers-Danlos Syndrome; Collagen Diseases | interventions — mecasermin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- mecasermin + Ehlers-Danlos (Active Comparator)
  Interventions: Drug: mecasermin
- Saline + Ehlers-Danlos (Placebo Comparator)
  Interventions: Drug: Saline
- Mecasamin + healthy control (Active Comparator)
  Interventions: Drug: mecasermin
- Saline + healthy control (Placebo Comparator)
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: mecasermin — 0,1 ml mecasermin (10 mg/ml) is injected intratendinous into the patella tendon with ultrasound guidance.
  Other Names: Increlex (mecasermin), Ipsen
  Arms: Mecasamin + healthy control; mecasermin + Ehlers-Danlos
Drug: Saline — 0,1 ml saline is injected intratendinous into the patella tendon with ultrasound guidance.
  Arms: Saline + Ehlers-Danlos; Saline + healthy control

SUMMARY:
The investigators want to inject insulin-like growth factor-I (IGF-I) into the patella tendon of Ehlers-Danlos patients and healthy controls to evaluate the response in collagen synthesis. Furthermore collagen synthesis is measured in muscle connective tissue and in skin.

The hypothesis is that the connective tissue in Ehlers-Danlos patients is more compliant and poorer in collagen than healthy controls, but that collagen synthesis can be stimulated by IGF-I.

DETAILED DESCRIPTION:
IGF-I will be injected with ultrasound guidance to one patella tendon and the other one will be injected with saline as control. Injections will be performed double blinded and timed 24 hours and 6 hours before tissue sampling.

Collagen synthesis will be measured as fractional synthesis rate based on stabile isotope technique using labelled proline.

10 patients diagnosed with Classical form of Ehlers-Danlos syndrome will be included and matched with 10 healthy controls based on age, gender, BMI and activity level.

The muscle biopsy will be taken from vastus lateralis muscle and the skin biopsy from the buttocks. The biopsies will if the size permits it also be used for histology and mRNA analyses.

ELIGIBILITY:
Inclusion Criteria:

* Classic form of Ehlers-Danlos syndrome OR healthy matched control

Exclusion Criteria:

* Malignity, cardiac diseases, diabetes, tendinopathy in patella tendons

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-09; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Fractional synthesis rate of collagen in tendon, muscle and skin | 6 hours
  A flood primed infusion of proline labelled with a stable isotope is used to calculate fractional synthesis rate of collagen in the 3 types of tissues. The infusion continues for 6 hours and tissue sampling is performed afterwards.

SECONDARY OUTCOMES:
Electron microscopy
  If there is additional tissue in the biopsies a piece will be stored for electron microscopy. In skin and tendon a transverse slice will be evaluated on collagen fibril diameter, form and density. In muscle the amount and appearance of connective tissue will be studied.
mRNA
  From the muscle biopsy a piece will be stored for mRNA analysis if possible. Targets will be collagen types and IGF-I isoforms.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kjaer, Professor, Study Director — Institute of Sportsmedicine Copenhagen
Locations (1):
- Institute of Sportsmedicine Copenhagen, Copenhagen, Denmark